CLINICAL TRIAL: NCT01288131
Title: Randomized Controlled Trial Study of Anti-r-HuEpo Associated PRCA Treated by Cyclosporine and Mycophenolate Mofetil (MMF) Compared With Cyclophosphamide and Prednisolone
Brief Title: Study of Anti-r-HuEpo Associated Pure Red Cell Aplasia (PRCA) Treatment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: We observed >90 % efficacy in cyclophosphamide and Prednisolone group for treatment of anti-i-HuEpo associated PRCA
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Kearkiat Praditpornsilpa, Associted Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/01_Medicine
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Anti-r-HuEpo Associated PRCA Subjects
Keywords: Anti-r-HuEpo antibody; Anti-r-HuEpo associated PRCA; Treatment; Absolute reticulocyte count
MeSH Terms: conditions — AIDS-Related Complex | interventions — Mycophenolic Acid; Cyclosporine; Cyclophosphamide; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSA+MMF (Active Comparator): Cyclosporine 100 mg BID combine with Mycophenolate mofetil 750 mg BID for 24 weeks
  Interventions: Drug: Cyclosporine combine with mycophenolate mofetil
- Cyclophosphamide + pred (Active Comparator): Cyclophosphamide 100 mg QD and prednisolone 1.0 mg/kg/day
  Interventions: Drug: Cyclophosphamide + pred

INTERVENTIONS:
Drug: Cyclosporine combine with mycophenolate mofetil — Cyclosporine 100 mg BID and mycophenolate mofetil 750 mg BID for 24 weeks
  Other Names: Neoral; Cellcept
  Arms: CSA+MMF
Drug: Cyclophosphamide + pred — Cyclophosphamide 100 mg QD combine with prednisolon 1.0 mg/kg/day
  Other Names: Endoxan
  Arms: Cyclophosphamide + pred

SUMMARY:
Recombinant human erythropoietin (r-HuEpo) has been used to treat renal anemia and improve morbidity and mortality in chronic kidney disease. Subcutaneous use of r-HuEpo causes immunogenicity and develops anti-r-HuEpo associated pure red cell aplasia (PRCA). The treatment of anti-r-HuEpo associated pure red cell aplasia is controversial. The investigators aim to evaluate the treatment for anti-r-HuEpo associated pure red cell aplasia in this study.

DETAILED DESCRIPTION:
Recombinant human erythropoietin was the first biotherapeutic medicinal product derived from recombinant DNA technology for the treatment of anemia in patients with chronic kidney disease (CKD). Although r-HuEpo raises hemoglobin levels in CKD and improves morbidity associated with anemia in CKD patients, the adverse immunological effect of r-HuEpo administered subcutaneously can result in anti-r-HuEpo associated PRCA. We aim to evaluate the effectiveness of two treatment protocol, cyclosporine combined with mycophenolate mofetil and cyclophosphamide combined with prednisolone for treatment of anti-r-HuEpo associated PRCA.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* CKD patient with anti-r-huEpo associated PRCA

Exclusion Criteria:

* Pregnancy or lactating women
* Receiving immunosuppression
* Active infection
* Previous history of allergic reaction to cyclosporine, mycophenolate mofetil, cyclophosphamide, prednisolone

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
anti-r-HuEpo antibody | Day 0 and month 6
  The anti-r-HuEpo antibody titer at day 0 (before treatment) and month 6 (6th month after treatment) of each arm will be compared

SECONDARY OUTCOMES:
Absolute reticulocyte count | Day 0 and month 6
  The Absolute reticulocyte count at day 0 (before treatment) and month 6 (6th month after treatment) of each arm will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Kearkiat Praditpornsilpa, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Kearkiat Praditpornsilpa, Bangkok, Thailand